CLINICAL TRIAL: NCT04105244
Title: Resourcefulness Intervention to Promote Self-Management in Parents of Technology-Dependent Children
Brief Title: Self-Management in Parents of Technology-Dependent Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Valerie Toly, Assistant Professor of Nursing, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20181088; R01NR017614 (NIH)
Record Dates: First submitted 2019-07-22; First posted 2019-09-26 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Caregivers; Parents; Self-Management; Chronic Illnesses, Multiple
Keywords: Mental Health; Physical Health; Technology-Dependent Children
MeSH Terms: conditions — Multiple Chronic Conditions; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The proposed study is a longitudinal (9-month) randomized controlled trial (RCT) in which primary caregiver parents of technology-dependent children will be randomly assigned to one of two study arms: (1) The Attention Control arm and (2) The Resourcefulness Training(c) arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data collectors and participants will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (No Intervention): The Attention Control arm will receive weekly phone calls for the first 4 weeks and at 2 and 4 months post-enrollment plus the current standard of care, whereby caregivers phone their healthcare providers when they have questions or concerns
- Resourcefulness Training Intervention© (Experimental): The Resourcefulness Training© arm will receive (a) individually tailored instruction on personal and social resourcefulness skills via the Resourcefulness Video and intervention nurse, (b) journal-writing instruction to describe resourcefulness application, (c) access to the study website with videotape vignettes and Resourcefulness Video, and (d) boosters at 2 and 4 months post-enrollment that will include reinforcement of skills learned and additional journal writing.
  Interventions: Behavioral: Resourcefulness Training©

INTERVENTIONS:
Behavioral: Resourcefulness Training© — The intervention includes self-help and help-seeking skills.
  Arms: Resourcefulness Training Intervention©

SUMMARY:
Parent caregivers of children with chronic conditions who require life-saving technology such as mechanical ventilation or feeding tubes must maintain a high level of vigilance 24 hours a day, 7 days a week. They usually provide a majority of their children's care and are often overwhelmed by the caregiving demands thus neglect health promotion behaviors that result in a deterioration of their own mental and physical health. The goal of this study is to test a cognitive-behavioral resourcefulness intervention that will improve these caregivers' mental and physical health and health promotion behaviors while they continue to provide vital care for these vulnerable children.

DETAILED DESCRIPTION:
Parent caregivers of children who require life-saving technology such as mechanical ventilation or feeding tubes must maintain a high level of vigilance 24 hours a day, 7 days a week. They report greater levels of stress, compromised self-management behaviors and poorer psychological and physical health than other caregiver groups which dramatically increases their mortality risk. Technology-dependent children (approximately 600,000) are among the sickest and most vulnerable subset of children with complex chronic conditions in the United States. They comprise 20% of all children discharged from the hospital to home, yet account for 61% of healthcare spending for children, up to $110 billion annually. Despite the adverse consequences for caregivers, there are no interventions to meet their specific needs. Resourcefulness Training, (cognitive-behavioral self-management intervention) has been shown to improve psychological and physical outcomes, mediate the effects of stress, and enhance the care provided to care-recipients. A Resourcefulness Training Intervention (RTI) will be tested in a randomized trial against an attention control group. The RTI includes face-to-face session for teaching social (help-seeking) and personal (self-help) resourcefulness skills, ongoing web access to the RTI video and video vignettes of caregivers of technology-dependent children describing resourcefulness skill application in daily life, 4 weeks of skills' reinforcement using daily log, weekly phone calls for the first 4 weeks, and booster sessions at 2 and 4 months post enrollment. The Attention Control group will receive weekly phone calls for the first 4 weeks and at 2 and 4 months post enrollment plus any usual care. The aims of the study are to: 1) Determine whether the RTI versus Attention Control improves psychological (mental HRQoL depressive cognitions, depressive symptoms, appraised stress, burden) and physical outcomes (physical HRQoL, chronic stress [hair cortisol]) over 9 months in parents of technology-dependent children, after controlling for covariates (parent race/ethnicity and gender, family income, and children's functional status, type of technology). 2) Determine whether changes in psychological and physical outcomes are mediated by changes in parents' levels of resourcefulness based on intervention condition. 3) Compare self-management behavior (sleep, positive health practices) over 9 months in parents who received RTI versus Attention Control. 4) Explore whether resourcefulness is a mediator between intervention condition and self-management behaviors controlling for baseline self-management behavior over 9 months. 5) Explore the relationship between self-management behavior and parent psychological and physical outcomes based on intervention condition. Our study will be the first to test a cognitive-behavioral RTI for this caregiver population. 6) Compare target children's ER visits, hospital days over 9 months based on parent intervention condition. If shown to be efficacious, it can be replicated with other caregivers of children with complex chronic conditions with strong potential for translation into practice.

ELIGIBILITY:
Inclusion Criteria:

* parent primary caregiver (biological, adoptive, or foster mother, father, grandmother, or grandfather) for a technology-dependent child based on the Office of Technology Assessment (OTA) classification criteria (Group 1, mechanical ventilators; Group 2, intravenous nutrition/medication; Group 3, respiratory or nutritional support);
* at least 18 years of age;
* able to speak and understand English;
* the technology-dependent child must be age 17.2 years or younger and receive care in the home from his/her parent. For children with more than one type of technology, we will follow OTA guidelines for classification.

Exclusion Criteria:

- Parents of children with a cancer diagnosis due to the short term use of technology following initial diagnosis and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A. Toly, PhD, RN, Principal Investigator — Frances Payne Bolton School of Nursing, Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Resource Sharing Plan: We support the principles, responsibilities and oversight of data sharing as articulated in the Final NIH Statement on Sharing Research Data (http://grants2.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). Once all data are collected, the research team will work to establish a database for the purpose of implementation of these standards, but with an emphasis upon the safeguarding of patient privacy, maintaining scientific integrity, and ensuring database privacy and security. Our goals will be to support the NIH intent of promoting dissemination of research findings and reagents to benefit NIH researchers country-wide and to promote rapid dissemination of clinical research findings. The data will be shared once all Human Subject identifiers are removed and preliminary analyses have been completed and collaborative ventures will be explored with the other investigators.
Supporting Information: SAP, CSR
Time Frame: The data will be shared once all Human Subject identifiers are removed and preliminary analyses have been completed and collaborative ventures will be explored with the other investigators.
Access Criteria: Must enter into data use agreement with Case Western Reserve University and the investigators.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 5 participants who signed the consent form but did not complete the baseline surveys and therefore they were not randomized and therefore not analyzed.
Groups:
- Resourcefulness Training Intervention©: The Resourcefulness Training© arm will receive (a) individually tailored instruction on personal and social resourcefulness skills via the Resourcefulness Video and intervention nurse, (b) journal-writing instruction to describe resourcefulness application, (c) access to the study website with videotape vignettes of caregivers of technology-dependent children describing resourcefulness skill application in daily life and Resourcefulness Video, and (d) boosters at 2 and 4 months post-enrollment that will include reinforcement of skills learned and additional journal writing.
  Resourcefulness Training©: Cognitive-behavioral intervention includes personal (self-help) and social (help-seeking) resourcefulness skills.
Period: Overall Study
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Started | 97 | 100
Completed | 67 | 62
Not Completed | 30 | 38
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Lost to Follow-up | 20 | 15
Not completed — Parent no longer eligible- child not living at home | 0 | 2
Not completed — Unable to contact to complete the intervention. | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | Resourcefulness Training Intervention© | Total
Number analyzed (Participants) | 97 | 100 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 95 | 97 | 192
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (9.58) | 35.9 (10.7) | 36.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 88 | 179
  Male | 6 | 12 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 90 | 93 | 183
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 18 | 16 | 34
  White | 71 | 77 | 148
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 97 | 100 | 197
Duration of Caregiving for Technology-Dependent Child [Mean (Standard Deviation); unit: months] — Number of months the parent has been caring for the child since they became dependent on medical technology.
  months | 43.3 (52.2) | 49.5 (47.4) | 46.3 (49.9)

OUTCOME MEASURES:

1. Primary Outcome: Psychological Outcome- Health Related Quality of Life
Description: Mental Health Related Quality of Life (The Patient-Reported Outcomes Measurement Information System [PROMIS] Short Form version 1.2- Global Health). Ten (10) Items. Score Range: 10 - 50. Global Mental Health (GMH) score converted to a T-Score metric - produces a physical and a mental health score. 10 points on the T-score metric is one standard deviation (SD). PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. A higher PROMIS T-score represents more of the concept being measured or better mental health.
Time Frame: Change Measured over 9 months of the study (baseline and 6 weeks, 3 months, 6 months, 9 months after baseline
Population: The number in the rows differs from the overall number analyzed because some of the participants withdrew or were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
score on a scale
  Baseline- Time 1: number analyzed (Participants) | 96 | 98
  Baseline- Time 1 | 40.5 (9.21) | 37.0 (8.85)
  6 weeks- Time 2: number analyzed (Participants) | 90 | 74
  6 weeks- Time 2 | 41.9 (8.95) | 39.70 (9.31)
  3 months- Time 3: number analyzed (Participants) | 81 | 71
  3 months- Time 3 | 41.7 (8.23) | 40.70 (9.04)
  6 months- Time 4: number analyzed (Participants) | 70 | 65
  6 months- Time 4 | 42.60 (9.41) | 41.00 (10.00)
  9 months- Time 5: number analyzed (Participants) | 62 | 60
  9 months- Time 5 | 42.40 (8.87) | 42.50 (8.61)
Statistical Analysis 1: Comparison: Attention Control vs Resourcefulness Training Intervention©; Test type: Superiority; p < 0.05, Mixed Models Analysis; Intent-to-treat principle using linear mixed-effects models with random intercepts to examine longitudinal change scores for the outcome; Wald tests = 0.05

2. Primary Outcome: Depressive Cognitions
Description: Screening Measure for Early Detection of Depressive Symptoms: The Depressive Cognition Scale. Measures depressive cognitions and negative thoughts that may lead to clinical depression. Eight (8) Items. Score Range: 0 - 40. Higher scores indicating more depressive cognitions.
Time Frame: Change Measured over 9 months of the study (baseline and 6 weeks, 3 months, 6 months, 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
score on a scale
  Baseline- Time 1 | 6.31 (5.09) | 8.27 (6.63)
  6 weeks- Time 2: number analyzed (Participants) | 90 | 74
  6 weeks- Time 2 | 6.93 (5.73) | 8.62 (6.27)
  3 months- Time 3: number analyzed (Participants) | 82 | 71
  3 months- Time 3 | 6.13 (2.08) | 8.17 (6.56)
  6 months- Time 4: number analyzed (Participants) | 70 | 65
  6 months- Time 4 | 5.84 (5.78) | 8.20 (7.32)
  9 months- Time 5: number analyzed (Participants) | 67 | 62
  9 months- Time 5 | 6.24 (6.06) | 6.69 (6.10)
Statistical Analysis 1: Comparison: Attention Control vs Resourcefulness Training Intervention©; Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Wald tests = .05

3. Primary Outcome: Physical Outcome
Description: (The Patient-Reported Outcomes Measurement Information System [PROMIS] Short Form version 1.2- Global Health). Ten (10) Items. Score Range: 10 - 50. Global Physical Health (GPH) score converted to a T-Score metric - produces a physical health score. 10 points on the T-score metric is one standard deviation (SD). PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population.
  Higher T-score means better physical health.
Time Frame: Change Measured over 9 months of the study (baseline and 6 weeks, 3 months, 6 months, 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
score on a scale
  Baseline- Time 1: number analyzed (Participants) | 96 | 98
  Baseline- Time 1 | 44.90 (7.58) | 44.00 (7.28)
  6 weeks- Time 2: number analyzed (Participants) | 90 | 74
  6 weeks- Time 2 | 46.00 (7.22) | 45.00 (8.07)
  3 months- Time 3: number analyzed (Participants) | 81 | 71
  3 months- Time 3 | 45.00 (7.31) | 46.10 (8.01)
  6 months- Time 4: number analyzed (Participants) | 70 | 65
  6 months- Time 4 | 45.10 (8.07) | 46.40 (8.53)
  9 months- Time 5: number analyzed (Participants) | 61 | 60
  9 months- Time 5 | 46.00 (7.23) | 48.20 (8.19)
Statistical Analysis 1: Comparison: Attention Control vs Resourcefulness Training Intervention©; Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Wald test = 0.05

4. Primary Outcome: Self-Management- Sleep- Subjective
Description: Appraised Sleep Quality (Pittsburgh Sleep Quality Index), Pittsburgh Sleep Quality Index The Pittsburgh Sleep Quality Index (PSQI). Assesses sleep quality and disturbances over a l-month time interval. Nineteen (19) items are grouped into seven component scores, each weighted equally on a 0-3 scale. Score Range (Global PSQI Score) is 0-21. Higher scores indicate worse sleep quality. Sub Scales are summed
Time Frame: Change Measured over 9 months of the study (baseline, 3 months, 6 months, 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
score on a scale
  Baseline- Time 1 | 7.134 (3.239) | 7.59 (2.903)
  3 months- Time 3: number analyzed (Participants) | 79 | 69
  3 months- Time 3 | 6.278 (3.4) | 6.768 (2.68)
  6 months- Time 4: number analyzed (Participants) | 69 | 64
  6 months- Time 4 | 6.058 (3.014) | 6.406 (2.866)
  9 months- Time 5: number analyzed (Participants) | 67 | 62
  9 months- Time 5 | 6.254 (2.93) | 6.161 (2.729)

5. Primary Outcome: Positive Health Practices
Description: Personal Lifestyle Questionnaire- Positive Health Practices Personal Lifestyle Questionnaire (PLQ). Measures the positive health practices of exercise, substance use, nutrition, relaxation, safety, and health promotion. Twenty-four (24) items 4-point summated rating scale with a range of possible scores from 24 to 96 Higher scores reflect the practice of more health behaviors. Total scores are reported.
Time Frame: Change Measured over 9 months of the study (baseline and 6 weeks, 3 months, 6 months, 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
score on a scale
  Female Baseline- Time 1: number analyzed (Participants) | 91 | 88
  Female Baseline- Time 1 | 64.515 (8.963) | 64.4 (8.357)
  Female 6 weeks- Time 2: number analyzed (Participants) | 84 | 63
  Female 6 weeks- Time 2 | 65.767 (9.054) | 65.811 (9.727)
  Female 3 months- Time 3: number analyzed (Participants) | 77 | 60
  Female 3 months- Time 3 | 66.805 (9.159) | 67.352 (8.626)
  Female 6 months- Time 4: number analyzed (Participants) | 64 | 55
  Female 6 months- Time 4 | 67.743 (8.421) | 68.277 (8.592)
  Female 9 months- Time 5: number analyzed (Participants) | 62 | 53
  Female 9 months- Time 5 | 66.642 (8.433) | 69.0 (9.987)
  Male Baseline- Time 1: number analyzed (Participants) | 6 | 12
  Male Baseline- Time 1 | 63.227 (8.433) | 63.35 (8.158)
  Male 6 weeks- Time 2: number analyzed (Participants) | 6 | 11
  Male 6 weeks- Time 2 | 64.233 (8.714) | 64.757 (9.379)
  Male 3 months- Time 3: number analyzed (Participants) | 5 | 11
  Male 3 months- Time 3 | 65.439 (8.844) | 66.254 (8.397)
  Male 6 months- Time 4: number analyzed (Participants) | 6 | 10
  Male 6 months- Time 4 | 66.329 (8.156) | 67.2 (8.337)
  Male 9 months- Time 5: number analyzed (Participants) | 5 | 9
  Male 9 months- Time 5 | 65.269 (8.288) | 67.597 (9.565)

6. Primary Outcome: Depressive Symptoms
Description: "Patient Reported Outcomes Measurement Information System (PROMIS)Short Form - Depressive Symptoms "Patient Reported Outcomes Measurement Information System (PROMIS)Short Form Version 1.0 - Depression 8a. Assess self-reported negative mood , views of self , social cognition, and decreased positive affect and engagement." Eight (8) Items. Score Range: 5 (Min)-40 (Max). Total Score is reported.
  The score is converted to a T-Score metric. 10 points on the T-score metric is one standard deviation (SD). PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. A higher PROMIS T-score represents more of the concept (depression) being measured thus a T-score of 60 is one standard deviation worse related to the concept of depression than average.
Time Frame: Change Measured over 9 months of the study (baseline and 6 weeks, 3 months, 6 months, 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
score on a scale
  Baseline- Time 1 | 51.80 (7.56) | 55.10 (7.87)
  6 weeks- Time 2: number analyzed (Participants) | 90 | 74
  6 weeks- Time 2 | 51.00 (7.53) | 53.10 (8.36)
  3 months- Time 3: number analyzed (Participants) | 82 | 71
  3 months- Time 3 | 50.10 (8.30) | 52.20 (8.11)
  6 months- Time 4: number analyzed (Participants) | 70 | 65
  6 months- Time 4 | 50.20 (8.45) | 50.90 (9.05)
  9 months- Time 5: number analyzed (Participants) | 67 | 62
  9 months- Time 5 | 49.90 (8.74) | 50.80 (7.86)
Statistical Analysis 1: Comparison: Attention Control vs Resourcefulness Training Intervention©; Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Wald test = 0.05

7. Secondary Outcome: Number of Technology-Dependent Children With ER Visits
Description: Number of Technology-Dependent Children with ER Visits over the time period the parent was enrolled and participating in the study from review of the children's charts.
Time Frame: Up to 9 months
Measure: Mean (Standard Deviation); unit: Number of ER visits
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
Number of ER visits | 0.9592 (1.566) | 0.9108 (1.569)
Statistical Analysis 1: Comparison: Attention Control vs Resourcefulness Training Intervention©; Test type: Superiority; p < 0.05, t-test, 2 sided

8. Secondary Outcome: Number of Technology-Dependent Children With Rehospitalizations
Description: Number of Technology-Dependent Children with Rehospitalizations over the time period the parent was enrolled and participating in the study from review of the children's charts.
Time Frame: Up to 9 months
Measure: Mean (Standard Deviation); unit: Number of rehospitalizations
Arm/Group | Attention Control | Resourcefulness Training Intervention©
Number analyzed (Participants) | 97 | 100
Number of rehospitalizations | 0.7755 (1.343) | 0.8415 (1.384)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Attention Control | Resourcefulness Training Intervention©
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/100
Other Adverse Events (participants affected / at risk) | 0/97 | 0/100

LIMITATIONS AND CAVEATS:
A majority of our study recruitment, enrollment, and data collection occurred during the Pandemic (2020-2021) therefore the protocol was modified to comply with the lockdown public health measures and the IRB mandate. All components of the study were conducted virtually using an institutional review board (IRB) approved videochat platform, REDCap, telephone, and text beginning in June 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT04105244/Prot_SAP_000.pdf